CLINICAL TRIAL: NCT02505776
Title: Safety and Patient Satisfaction With GLASH VISTA™ (Bimatoprost 0.03%) in the Treatment of Eyelash Hypotrichosis in Japan
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 192024-089
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GLASH VISTA™: Patients with eyelash hypotrichosis prescribed bimatoprost cutaneous solution 0.03% (GLASH VISTA™) as per local standard of care in clinical practice.
  Interventions: Drug: Bimatoprost cutaneous solution 0.03%

INTERVENTIONS:
Drug: Bimatoprost cutaneous solution 0.03% — Bimatoprost cutaneous solution 0.03% (GLASH VISTA™) prescribed as per standard of care in clinical practice.
  Other Names: GLASH VISTA™; Latisse®

SUMMARY:
This is a post-marketing surveillance study in Japan that will evaluate the safety and patient satisfaction with GLASH VISTA™ (bimatoprost cutaneous solution 0.03%) in the treatment of hypotrichosis of the eyelashes.

ELIGIBILITY:
Inclusion Criteria:

-Patients who have been prescribed GLASH VISTA™ in clinical settings and filled at least one prescription for GLASH VISTA™.

Exclusion Criteria:

-None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eyelash hypotrichosis
Sampling Method: Non-Probability Sample
Enrollment: 1699 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to 12 Months
Change from Baseline in Patient Satisfaction with Eyelashes As Measured by the 3-Item Patient Eyelash Satisfaction Survey | Baseline, Month 1
Change from Baseline in Patient Satisfaction with Eyelashes As Measured by the 3-Item Patient Eyelash Satisfaction Survey | Baseline, Month 4
Change from Baseline in Patient Satisfaction with Eyelashes As Measured by the 3-Item Patient Eyelash Satisfaction Survey | Baseline, Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne St. Rose, Dr, Study Director — Allergan
Locations (1):
- Tokyo, Japan

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com